CLINICAL TRIAL: NCT02675595
Title: Prospective Evaluation of Fetal Intelligent Navigation Echocardiography (FINE)(5D) Versus Conventional 2D Echocardiography in Comprehensive Fetal Cardiac Imaging in the Second Trimester of Pregnancy
Brief Title: 5D Versus Conventional 2D Fetal Echocardiography During Second Trimester of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omneya Nagy ELmakhzangy, Specialist, Ain Shams University
Other Study IDs: MD thesis
Record Dates: First submitted 2016-01-21; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis:

In Women in the second trimester of pregnancy 5D offers an alternative method for fetal Echocardiography compared to conventional 2D scanning

Question:

Does 5D software technology is as efficient as 2D scanning in fetal echocardiography of second trimesteric fetuses?

Aim:

This study aims at assessing the accuracy of performance of the 5D as a new scanning technology in fetal Echocardiography compared to the conventional use of 2D scanning.

DETAILED DESCRIPTION:
Congenital malformations account for more than 20% of all infant deaths(CDC,2014), and congenital heart defects are the most common types of birth defects.

The prenatal diagnosis of major congenital heart defects remains a challenge. Publications by Acherman et al (Acherman RJ .et al) and Sklansky et al (Sklansky MS.et al)have found that approximately 35% of cardiac anomalies are detected prenatally, a frequency that is not substantially different from that documented by Wigton et al in 1993 (Wigton TR, et al) Advances in prenatal ultrasonography have improved prenatal care in recent decades and increased the detection of a large number of congenital malformations. The prenatal detection rate of congenital heart disease (CHD), however, has not shown the same increase as the detection of malformations in other fetal systems (DeVore GR, et al). CHDs are the most commonly overlooked lesions in prenatal screening programs(Garne E et al, Tegnander E et al). This causes concern as CHD represents the most common congenital malformation and is the leading cause of infant mortality in the first year of postnatal life(Garne E). It has been estimated that the prevalence of CHD is 4-8 per 1000 neonates(Hoffman JI et al).

Early detection and accurate prenatal diagnosis of CHD reduces neonatal morbidity and mortality rates by allowing provision of adequate prenatal and postnatal care(Randall P et al, Goncalves LF et al). Before viability is reached, parents can be counseled on the diagnosis, severity and prognosis. Furthermore, it provides parents with the opportunityto make informed decisions on the further course of pregnancy. The four-chamber view has become the standard approach in screening for CHD. Identification of the right and left outflow tracts markedly improves the detection rate of CHD(DeVore GR et al, Stumpflen I et al).

Prenatal detection of these anomalies has proved challenging. In a British study from 1999, Bull(AIUM 2013) reported on 4799 pregnancies affected by major congenital heart defects and found that the antenatal detection rate was only 24%. Lower detection rates were noted in centers that only assessed the 4-chamber view. Correspondingly, in an attempt to improve the antenatal detection rates of congenital heart defects, the American Institute of Ultrasound in Medicine, American College of Obstetricians and Gynecologists, and International Society of Ultrasound in Obstetrics and Gynecology all have recommended that an attempt should be made to image the ventricular outflow tracts during the fetal anatomic survey.( Carvalho JS et al. , Bull C., AIUM 2003)

However, imaging of these outflow tracts can be challenging, and it is not clear that they can be typically obtained in generalized non-tertiary care settings. A 2007 study from the United States, which included 77,000 births, found that only 36% of major congenital heart defects were detected antenatally. It is not clear from the study whether outflow views were routinely obtained at all of the laboratories involved, but the study suggests that better detection rates could be achieved if outflow views were more routinely imaged.( Bull C. )

In an effort to improve antenatal detection of these anomalies, the American Institute of Ultrasound in Medicine, the American College of Obstetricians and Gynecologists, and the International Society of Ultrasound in Obstetrics and Gynecology have suggested that routine ultrasound examinations should attempt to include views of the cardiac outflow tracts. (AIUM 2003)

The myriad of fetal positions and the different maternal factors that influence the examination make fetal echocardiography one of the more difficult tasks for sonographers. To help improve and standardize fetal cardiac examinations, Yagel et al. and Yoo et al. described a method in which five cardiac planes are visualizedfor a complete examination of the fetal heart(Yoo SJ et al,Yagel et al ). Additionally, three- and four-dimensional (3D and 4D) ultrasound imaging can be a valuable tool in fetal echocardiography(ACOG 2004, Chaoui R et al,AIUM 2010, Yagel S et al M. C. Haak et al , Luciane Alves Rocha et al Rocha LA et al )

Other proposals have included obtaining routine 2-dimensional (2D) cine clips, universal fetal echocardiography, and routine use of 3-dimensional (3D) fast acquisition volumes. One reason that 3D sonographic technologies have been suggested is because routine visualization of cardiac views has proven to be a challenge with 2D imaging in centers that are less experienced with prenatal diagnosis, and 3D stored volumes could then be evaluated further by those more experienced.( M. C. Haak et al , Luciane Alves Rocha, et al, Rocha LA et al )

Fetal Intelligent Navigation Echocardiography (FINE) 5D work flow refers to semi-automated identification of specific diagnostic image planes and measurements from a volume dataset simultaneously displaying nine standard fetal cardiac views. It allows the examination of cardiac planes, such as the axial planes and view of the interventricular septum (IVS plane) which are technically very difficult to image using conventional two-dimensional (2D) echocardiography (Rocha LA et al).

However, to be an effective tool in fetal echocardiography, 5D volume acquisition must be feasible in routine clinical practice. A number of reports on these new technologies have emphasized the requirement of a substantial learning curve for the use of 5D ultrasound imaging(M. C. Haak et al , Luciane Alves Rocha et al ). This may explain the delay in widespread introduction of this new technique in first- and second level ultrasound departments, and even in tertiary referral centers.

ELIGIBILITY:
Inclusion Criteria:

* Living fetus.
* Singleton
* No gross fetal structural malformation
* No maternal Medical Disorders
* G.A : in between 20-26 wks.
* Verbal consent informing the aim and process of this study

Exclusion Criteria:

* the fetal spine between the 9- and 3-o'clock positions
* Missed Abortion.
* women with body mass index (BMI) ≥30 kg/m2
* GA : before 20 wk.
* presence of polyhydramnios or oligohydramnios (amniotic fluid index >95th percentile or < 5th percentile)
* Detectable or suspected fetal cardiac anomaly
* Fetal congenital malformation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Second trimester pregnant women
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Obtaining standard 9 views of fetal echocardiography by 5D as well as 2D | 2 years
  All 80 fetuses will undergo 2D and 5D detailed fetal echocardiography to obtain the standard nine cardiac views according to standards set by AIUM (American Institute of Ultrasound in Medicine) and both modalities will be compared by their ability to obtain the nine standard cardiac views.

CONTACTS AND LOCATIONS:
Overall Officials: Omneya Nagy ELmakhzangy, masters, Principal Investigator — Specialist at Ain Shams University; Omneya Nagy ELmakhzangy, masters, Principal Investigator — Specialist Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided